CLINICAL TRIAL: NCT00182013
Title: Open-Label Comparative Study of Risperidone Versus Olanzapine Versus Quetiapine for Mania in Children and Adolescents With Bipolar I and Bipolar II Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001P-000259
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Bipolar Spectrum Disorder
MeSH Terms: interventions — Risperidone; Olanzapine; Quetiapine Fumarate

INTERVENTIONS:
Drug: Risperidone — Open treatment with Risperidone
Drug: Olanzapine — Open treatment with Olanzapine
Drug: Quetiapine — Open treatment with Quetiapine

SUMMARY:
The objective of this study is to compare the safety and effectiveness of Risperidone, Olanzapine, and Quetiapine in the treatment of mania in children and adolescents with Bipolar disorder over 8 weeks and then over an extension phase. This is an exploratory, open-label study, which seeks to determine if there is evidence for efficacy. The results of this study will be used to generate hypotheses for a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 6 to 18 years of age
* Patient must have a diagnosis of bipolar I or bipolar II disorder and currently displaying an acute manic, hypomanic, or mixed episode (with or without psychotic features) according to the DSM-IV based on clinical assessment and confirmed by structured diagnostic interview (Kidd Schedule of Affective Disorders).
* Patients must have an initial score on the Y-MRS total score of at least 15.
* Patient must be able to participate in mandatory blood draws.
* Patient must be able to swallow pills.

Exclusion Criteria:

* Patients with chronic medical illness, DSM-IV substance dependence within the past 6 months, pregnant or nursing females, and those at serious risk of suicide will be excluded from the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2001-06; Primary Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Young Mania Rating Scale | baseline to 8 weeks
  Improvement defined as score reduction of 30% or greater.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — MGH

REFERENCES:
- [Derived] Joshi G, Petty C, Wozniak J, Faraone SV, Doyle R, Georgiopoulos A, Hammerness P, Walls S, Glaeser B, Brethel K, Yorks D, Biederman J. A prospective open-label trial of quetiapine monotherapy in preschool and school age children with bipolar spectrum disorder. J Affect Disord. 2012 Feb;136(3):1143-53. doi: 10.1016/j.jad.2011.09.042. Epub 2011 Oct 28. PMID 22035648